CLINICAL TRIAL: NCT06595030
Title: Methodology Issues in a Tailored Light Treatment for Persons With Dementia - Aim 3
Brief Title: Investigating the Impact of Duration and Amount of Light on the Circadian System Response - Aim 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-20-01736 Aim 3; 5R01AG034157-13 (NIH)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Lighting Intervention (Active Comparator): Combining spectrum and light level, the active TLI will allow the researchers to use a light source that will stimulate the circadian system and provide the participants with options as to how the light treatment will be delivered.
  Interventions: Device: Active Lighting Intervention
- Control Lighting Intervention (Placebo Comparator): The control TLI will allow the researchers to use a light source that will not stimulate the circadian system and provide the participants with options as to how the light treatment will be delivered.
  Interventions: Device: Control Lighting Intervention

INTERVENTIONS:
Device: Active Lighting Intervention — The TLI will allow researchers to use a light source that will control how the circadian system is stimulated and provide the participants with options as to how the light treatment will be delivered.
  Other Names: TLI
  Arms: Active Lighting Intervention
Device: Control Lighting Intervention — The TLI will allow researchers to use a light source that will not stimulate the circadian system and provide the participants with options as to how the light treatment will be delivered.
  Other Names: TLI
  Arms: Control Lighting Intervention

SUMMARY:
Investigate the long-term impact of amount and duration of Tailored Lighting Intervention (TLI) obtained from Aims 1 and 2 on sleep, cognition, circadian marker, mood, and behavior in AD/ADRD patients. For this single-arm, randomized, placebo-controlled study, the researchers plan to recruit 100 participants who will experience either the active TLI or the placebo for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease or related dementia with a Montreal Cognitive Assessment score <25
* Sleep disturbance with a Pittsburgh Sleep Quality Index score ≥5

Exclusion Criteria:

* Extensive brain vascular disease, traumatic brain injury, multiple sclerosis, Parkinson's Disease
* Obstructing cataracts
* Severe macular degeneration
* Use of sleep medication
* Use of oral melatonin
* untreated moderate to severe sleep apnea
* Severe restless leg syndrome - Blindness

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Disturbance using the Pittsburgh Sleep Quality Index (PSQI) | Up to Week 36
  The PSQI is used to measure sleep quality and is composed of 19 items that generate 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each subscale is scored 0 to 3. The sum of the 7 component scores yields a single global score with a full scale range of 0 to 21. A higher score indicates higher sleep disturbance.

SECONDARY OUTCOMES:
Sleep efficiency using actigraphy | Up to Week 36
  Actigraphs will be worn continuously for 7 days during each assessment week. Changes in sleep efficiency will be measured using the actigraphy software. Sleep efficiency is a calculated as a ratio of the time spent in bed and the time spent sleeping
Depression using the Cornell Scale for Depression in Dementia (CSDD) | Up to Week 36
  The CSDD is a 19-item tool designed to rate symptoms of depression in patients with dementia. Full Scale ranges from 0 to 38 with a higher score indicating greater depression.
Agitation using the Cohen-Mansfield Agitation Inventory (CMAI) | Up to Week 36
  The CMAI assesses the frequency of manifestations of agitated behaviors in elderly persons. The CMAI is a caregivers' rating questionnaire consisting of 29 agitated behaviors, each rated on a 7-point scale of frequency. Score ranges from 30 to 210 with a higher score indicating higher agitated behavior.
Light measurements using the Daysimeter | Up to Week 36
  Circadian light measurements will be collected during waking hours for 7 days each assessment week using the daysimeter. The light measurement is reported as Lux levels.
Cognitive status Using the Montreal Cognitive Assessment (MOCA) | Up to Week 36
  The MoCA is a 1-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. Total score range from 0 to 30. Lower score indicates lower cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, Menands, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared not individual